CLINICAL TRIAL: NCT00758225
Title: A Phase II Open-label Extension Study to Obtain Long-term Safety, Tolerability and Efficacy Data of Idebenone in the Treatment of Duchenne Muscular Dystrophy - Extension to Study SNT-II-001
Brief Title: Long-term Safety, Tolerability and Efficacy of Idebenone in Duchenne Muscular Dystrophy (DELPHI Extension)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Thomas Meier, PhD / Chief Scientific Officer, Santhera Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN T-II-001-E
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Duchenne; Idebenone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — idebenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- only one arm (Experimental)
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone — Patients ≤ 45 kg: 450 mg/day (1 tablet 3 times a day) Patients > 45 kg: 900 mg/day (2 tablets 3 times a day)

SUMMARY:
The scientific aim of the present extension study is to monitor long-term safety and tolerability of idebenone in patients with DMD. Furthermore, the long-term effect on respiratory, cardiac and motor functions, and skeletal muscle strength/function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study SNT-II-001
* Body weight ≥ 25 kg
* Glucocorticosteroids and ACE-inhibitors are allowed, if on stable dosage within 2 months prior to inclusion
* Eligibility to participate in the present extension study as confirmed by the investigator

Exclusion Criteria:

* Safety or tolerability issues arising during the course of SNT-II-001 which in the opinion of the investigator preclude further treatment with idebenone
* Clinically significant abnormalities of haematology or biochemistry
* Abuse of drugs or alcohol
* Use of coenzyme Q10 or idebenone within 30 days prior to inclusion
* Intake of any investigational drug within 30 days prior to inclusion
* Symptomatic heart failure
* Previous history of ventricular arrhythmias (other than isolated ventricular extrasystole); ventricular arrhythmias presented at baseline
* Known individual hypersensitivity to idebenone or to any of the excipients

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Measures of safety and tolerability of idebenone: - Nature and frequency of AEs - Laboratory parameters (haematology, biochemistry and urinalysis) - Physical examinations and vital signs - ECGs | Month 0, 3, 6, 12, 18, 24, FU

SECONDARY OUTCOMES:
Measures of efficacy of idebenone: - Respiratory Function Testing - Motor Function Measure - Quantitative Muscle Testing - Hand-Held Myometry - Echocardiography and Color Doppler Myocardial Imaging - Cardiac biomarkers | Month 0, 6, 12, 18, 24

CONTACTS AND LOCATIONS:
Overall Officials: Prof Gunnar Buyse, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium